CLINICAL TRIAL: NCT04911569
Title: The Effect of Ultrasound-guided Cryoneurolysis on Persistent Cutaneous Neuropathic Pain After Surgery and Trauma
Brief Title: Cryoneurolysis for Cutaneous Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cryo_210510_V02
Record Dates: First submitted 2021-05-19; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Non-blinded, non-randomized, non-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoneurolysis (Experimental): All 25 patients will receive cryoneurolysis
  Interventions: Device: Cryoneurolysis

INTERVENTIONS:
Device: Cryoneurolysis — Cryoneurolysis

SUMMARY:
Feasibility study with 25 patients investigating the effect of cryoneurolysis on persistent cutaneous neuropathic pain after surgery and trauma. All patients receive active treatment (cryoneurolysis). The study design is unblinded, non-randomized, non-controlled.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* ASA (American Society of Anesthesiologists) physical status classification system I-III
* Informed consent
* Capable of subjective evaluation of pain
* Capable of reading and understanding Danish and informed written consent
* Average pain intensity >49/100 on VAS in the primary focal pain area for a minimum of 6 months at the time of inclusion
* Relevant injury (surgery or trauma) of peripheral nerves
* Plausible cutaneous location of pain
* In the area of pain, at least one of the following (1-8): (1) Hypo/anesthesia for touch/brush (2) Hypo/anesthesia for cold (3) Hypo/anesthesia for warmth (4) Hypo/anesthesia for pinprick (5) Allodynia for touch/brush (6) Allodynia for cold (7) Allodynia for warmth (8) Hyperalgesia for pinprick
* Neuropathic pain score (Douleur Neuropathique en 4 Questions, DN-4) >3/10
* Definitive diagnosis of neuropathic pain (Finnerup et al 2016)

Exclusion Criteria:

* Inability to cooperate
* Inability to understand Danish
* Allergy to local anesthetic
* Infection in the area of cryo probe insertion
* Significant competitive chronic pain
* Progressive neurologic disease
* Increased risk at needle insertion and cold exposure (e.g. Raynaud, coagulopathies)
* Uncontrolled severe systemic disease
* Implanted electronic devices unless approved by the relevant medical specialist
* Previous cryoneurolysis with no relevant effect for the same neuropathic pain
* Previous interventional pain therapy (e.g. spinal cord stimulation) with no relevant effect for the same neuropathic pain
* Expected duration of life < 2 years
* Pregnancy
* Abuse of alcohol, narcotics or medicine
* Current psychiatric disease
* Inclusion in other clinical trials
* Ongoing patient complaint
* Body mass index < 18.5 or > 34.9 kg/m2
* Change of pain therapy within the last 28 days prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-07 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Success of cryoneurolysis | 1 hour after cryoneurolysis
  Frequency of patients with > 50% reduction of neuropathic pain

SECONDARY OUTCOMES:
Axonal loss estimated before cryoneurolysis | Maximum one year prior to the cryoneurolysis procedure
Hyperalgesia for pinprick | 1 hour after cryo procedure compared to baseline
  Visual Analogue Scale (VAS) score (0-100)
Allodynia for brush | 1 hour after cryo procedure compared to baseline
  VAS score (0-100)
Frequency of NRS score < 4 | 1 hour, 2 weeks and 1,2,3,4,5 and 6 months after cryo procedure
  Numeric Rating Scale (NRS) score (0-10)
Pain score | 1 hour, 2 weeks and 1,2,3,4,5 and 6 months after cryoneurolysis procedure
  NRS score (0-10)
Duration of freedom of pain (number of days after the cryoneurolysis procedure) | Maximum follow-up until 12 months after cryoneurolysis procedure
  NRS < 4
Change of neuropathic pain score DN-4 | 1 hour, 2 weeks and 1,2,3,4,5 and 6 months after cryo procedure
  DN-4 = Douleur Neuropathique en 4 Questions
Patient satisfaction at completion of cryo procedure | From skin insertion of cryo probe to withdrawal of cryo probe
  NRS score (0-10)
Change in muscle strength of relevant muscle groups | 1 hour after cryoneurolysis compared to baseline
  Handheld dynamometer
Procedure time for cryoneurolysis | From skin insertion of cryo probe to withdrawal of cryo probe
Pain related medication | 2 weeks and 1,2,3,4,5 and 6 months after cryo procedure
PGIC | 2 weeks and 1,2,3,4,5 and 6 months after cryo procedure
  Patient Global Impression of Change
Adverse events | 1 hour, 2 weeks and 1,2,3,4,5 and 6 months after cryo procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Bendtsen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No